CLINICAL TRIAL: NCT03257033
Title: Targeted Intra-arterial Gemcitabine vs. Continuation of IV Gemcitabine Plus Nab-Paclitaxel Following Induction With Sequential IV Gemcitabine Plus Nab-Paclitaxel and Radiotherapy for Locally Advanced Pancreatic Cancer
Brief Title: Intra-arterial Gemcitabine vs. IV Gemcitabine and Nab-Paclitaxel Following Radiotherapy for LAPC
Acronym: TIGeR-PaC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RenovoRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RR3 [CP-03-001]
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Subjects with stable or responding disease after approximately four months of induction therapy, and who are not surgical candidates will then be randomized to be in either the test group or control group. Crossovers are not allowed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IA Therapy (Experimental): IA Treatments with 1,000 mg/m2 gemcitabine administered through RenovoCath every other week for a maximum of 8 treatments for approximately 16 weeks.
  Interventions: Drug: Gemcitabine; Device: RenovoCath
- IV Therapy (Active Comparator): IV gemcitabine and nab-paclitaxel will be administered for 16 weeks on days 1, 8, and 15 of a 28 day cycle. Nab-paclitaxel will be administered intravenously following pre-medication at a dose of 125 mg/m2 over 30 minutes followed by an infusion of gemcitabine at a dose of 1000 mg/m2 over 30 minutes.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Chemotherapy
  Other Names: Gemzar
Drug: nab-paclitaxel — Chemotherapy
  Other Names: Abraxane
  Arms: IV Therapy
Device: RenovoCath — Intra-arterial catheter
  Arms: IA Therapy

SUMMARY:
The study is a multi-center, open-label, randomized active controlled study of subjects with locally advanced pancreatic adenocarcinoma which is unresectable.

DETAILED DESCRIPTION:
All subjects will receive induction therapy of IV gemcitabine plus nab-paclitaxel, as well as SBRT radiation therapy for approximately a total of four months. Subjects who remain eligible will then be randomized to receive either intra-arterial chemotherapy with gemcitabine; or to continue gemcitabine plus nab-paclitaxel. Subjects will receive the randomized treatments for up to 16 weeks or until progression. Both groups will receive either IV gemcitabine and nab-paclitaxel or oral capecitabine following the 16-week treatment course until disease progression at the discretion of the Investigator and then followed for survival for five years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or Cytopathology confirmed pancreatic adenocarcinoma with initial diagnosis within 8 weeks of consent for patients who enroll at cycle 1, and from the start of cycle 1 of gemcitabine + nab-paclitaxel chemotherapy for patients who enroll at cycle 2
2. Locally advanced, unresectable disease at screening and prior to randomization, as defined by NCCN criteria determined by an on-site, experienced, multidisciplinary team (as confirmed by CT or MRI within 30 days of the start of cycle 1)
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
4. Age ≥ 18 years
5. Adequate laboratory values prior to receiving the first dose of nab-paclitaxel and gemcitabine: (criterion must be met prior to cycle 2.) For a subject with elevated bilirubin, AST or ALT, who has had a biliary stent placed, if the subject's lab values have returned to within the required range for eligibility noted below in sub-criteria e and f [(AST) ALT ≤ 3.0 X the upper normal limit, and total bilirubin ≤ 1.5 X the upper normal limit] after placement of stent and prior to cycle 2, he/she is eligible for the study. Additional details regarding eligibility for subjects who have had biliary stents recently placed are outlined in sub-criteria f and h below.

   1. Absolute neutrophil count (ANC) ≥ 1,500/μL
   2. Platelet count ≥ 100,000/μL
   3. Hemoglobin ≥ 9.0 g/dL
   4. Serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine >1.5 mg/dL
   5. *Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 X the upper normal limit of institution's normal range
   6. *Total bilirubin ≤ 1.5 X the upper normal limit of institution's normal range -OR- If biliary stent is placed or planned to be placed within 6 weeks of Cycle 1 Day 1 (C1D1), total bilirubin ≤ 2.0 X the upper normal limit of institution's normal range (see section 9.1.4 for dose modification due to elevated bilirubin)
   7. Prothrombin time (PT) and partial thromboplastin time (PTT) must be ≤ 1.5 X upper normal limit of institution's normal range. Subjects who are currently taking anti-coagulant therapy are eligible if not meeting this criterion
   8. International normalized ration (INR) ≤ 1.5 X upper normal limit of institution's normal range. Subjects who are currently taking anti-coagulant therapy are eligible if not meeting this criterion *For elevated AST, ALT, and total bilirubin at screening, subject must have a normalized result prior to initiation of Cycle 2 if abnormal labs are considered related to bile duct obstruction and a biliary stent has been placed
6. Life expectancy > 12 weeks
7. Negative pregnancy test for women of childbearing potential (either serum or urine) within one day prior to administration of the first dose of chemotherapy. Women of childbearing potential should use highly effective methods of contraception during treatment and for up to 6 months following treatment cessation
8. Provide written informed consent
9. Subjects willing to participate in the study for at least 8 months if randomized to IA gemcitabine OR IV gemcitabine + nab-paclitaxel

Exclusion Criteria:

1. Any prior treatment for pancreatic cancer OR more than one cycle of gemcitabine and nab-paclitaxel treatment. For subjects who have started on their first cycle of gemcitabine and nab-paclitaxel treatment prior to consent, Inclusion Criterion #1 only applies to the first gemcitabine and nab-paclitaxel dose and must be within 6 weeks of confirmed diagnosis
2. Any evidence of metastatic disease or another active malignancy within the past one year except for cervical cancer in situ, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin.
3. Subjects unable or unwilling to have their first randomized treatment within 3 weeks of the post induction imaging and within 5 weeks of their last induction treatment
4. Subjects without baseline tumor imaging
5. As determined by the Sponsor:

   Arterial anatomy unsuitable for IA delivery of gemcitabine to the intended tumor site, determined by CT or MRI, as determined and approved by the Sponsor Imaging Advisor, which includes the following:
   1. Stenosis or occlusion in the intended artery for treatment
   2. Inability to exclude major side branches in the area of the intended RenovoCath® catheter occlusion
   3. No suitable artery with a diameter greater than 3 mm in proximity of at least one side of the tumor
   4. Superior mesenteric vein (SMV) occlusion or stenosis that cannot be resolved with medication or intervention prior to randomization, if the superior mesenteric artery (SMA) is the only viable treatment artery Note: Arterial Anatomy will be reviewed by the Sponsor, RenovoRx Imaging Advisor, and RenovoRx Medical Monitor for approval
6. Contraindications for SBRT planning which includes the following:

   1. Gastrointestinal mucosal infiltration evident at the time of diagnostic endoscopy
   2. Prior abdominal radiotherapy judged to have clinically significant degree of overlap with planned SBRT dose distribution Note: Primary tumors with a diameter greater than 7 cm must be assessed on a case-by-case basis with the RenovoRx Imaging Advisor prior to excluding the subject from the trial.
7. Subjects with known HIV infection or active viral hepatitis
8. Severe infections requiring hospitalization within 4 weeks prior to the first study treatment, including but not limited to complications of infection, bacteremia or severe pneumonia
9. Signs or symptoms of infection within 2 weeks prior to the first study treatment, as assessed by the Investigator
10. Received antibiotics for treatment of an infection within 48 hours prior to initiation of study treatment. Subjects receiving prophylactic antibiotics are eligible
11. History of severe allergic, anaphylactic, or other hypersensitivity reactions to gemcitabine or nab-paclitaxel
12. Any anti-cancer therapy including chemotherapy, hormonal therapy for prostate cancer, or radiotherapy within 2 weeks prior to initiation of study treatment; or herbal therapy intended as anti-cancer therapy within 1 week prior to initiation of study treatment
13. Subjects with uncontrolled seizures
14. Cardiovascular disease including unstable angina or life-threatening cardiac arrhythmia, myocardial infarction, stroke; or New York Heart Association (NYHA) Class III or IV congestive heart failure (CHF) within the last 3 months prior to the first study treatment. Subjects with prior history of Myocardial Infarction (MI), congestive heart failure (CHF), coronary artery bypass grafting, or prior valve surgery need to have assessment of ejection fraction (EF) to ensure EF is not ≤ 40% (as determined by MRI, ECHO, or Nuclear Scan), within the last 3 months prior to the initiation of study treatment
15. Other severe concurrent disease or comorbidities which make it difficult to participate in this study, as assessed by Investigator
16. Any of the following procedures prior to initiation of study treatment:

    1. Catheterization, endoscopy, stent or drain placement within 48 hours. (Diagnostic laparoscopy without surgical intervention and/or port placement do not require any wait time prior to study treatment)
    2. Minor surgery requiring light sedation (such as surgical laparoscopy) within 2 weeks
    3. Major surgery within 4 weeks
17. Women who are breastfeeding
18. Male or female subjects of reproductive potential who do not agree to either remain abstinent or employ highly effective and acceptable forms of contraception throughout their participation in the study and for 6 months after the last study treatment
19. Subjects receiving any other investigational agents within 2 weeks prior to the initiation of treatment
20. Any social situations or psychiatric illness that would limit compliance with study requirements
21. Subjects unable or unwilling to have standard catheterization procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2018-03-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to Five Years
  OS from time of randomization will be calculated using the Kaplan-Meier method and compared between the test and control groups using the stratified Wilcoxin Test

SECONDARY OUTCOMES:
Overall Survival for treatment received and unresected populations | Up to Five Years
  The primary endpoint analysis will be repeated for the Treatment Received and Unresected Subject populations.
Progression Free Survival | Up to Five Years
  To compare the Progression Free Survival of intra-arterial delivery of gemcitabine using the RenovoCath™ device vs. continuation of IV gemcitabine and nab-paclitaxel following induction therapy with gemcitabine and nab-paclitaxel and radiation treatment for locally advanced pancreatic adenocarcinoma. Disease response and progression will be assessed according to RECIST 1.1.
Objective response rate and duration of response | Up to Five Years
  Objective response is defined as a complete response, CR, or partial response, PR, determined by Investigator assessment and confirmed by repeat assessment ≥ 4 weeks after initial documentation.
Health Related Quality of Life | Up to Five Years
  The EORTC questionnaire will be used to assess health related quality of life. The summary scores for the EORTC questionnaire will be calculated at baseline and follow-up.
Neuropathy Assessment | 1 Year
  The degree of neuropathy will be measured by the FACT/GOG-NTX-4 (version 4). The results will be cross tabulated by randomized treatment group for each study visit.
Frequency of neutropenia | 30 Days Post-Randomized Treatment
  Neutropenia with onset after randomization requiring the use of filgrastim or other medications for white blood cell stimulation will be compared between the test and control groups through progression of disease.
Frequency of Myelosuppression | 30 Days Post-Randomized Treatment
  Frequency of myelosuppression requiring medication for blood products to overcome anemia, neutropenia, and thrombocytopenia
Safety, defined as adverse event rate, and tolerability, defined as occurrence of treatment discontinuation | Up to Five Years
  Safety and tolerability of the drug/device combination will be assessed by the occurrence of treatment discontinuation and the presence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Pishvaian, Study Chair — Johns Hopkins Kimmel Cancer Center
Locations (42):
- United States (36):
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Sutter Cancer Center Sacramento, Sacramento, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado, CCCRIC, Englewood, Colorado
  - Sibley Memorial Hospital - a member of Johns Hopkins medicine, Washington D.C., District of Columbia
  - Georgetown University, Washington D.C., District of Columbia
  - 21st Century Oncology, Fort Myers, Florida
  - Miami Cancer Center, Miami, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - ASCLEPES Research Centers, Weeki Wachee, Florida
  - Piedmont-Columbus Regional - John B. Amos Cancer Center, Columbus, Georgia
  - University of Iowa Hospitals and Clinics - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - LSU Health Shreveport, Shreveport, Louisiana
  - Medstar Franklin Square, Baltimore, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - MD Anderson Cancer Center at Cooper Hospital, Camden, New Jersey
  - Atlantic Health System - Morristown Medical Center, Morristown, New Jersey
  - Albany Stratton VA Medical Center, Albany, New York
  - Feinstein Institutes for Medical Research - Northwell Health, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Hospital, The Bronx, New York
  - Levine Cancer Institute - Atrium Health, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Oklahoma University - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina - Hollings Cancer Center, Charleston, South Carolina
  - Prisma Health (formerly Greenville Health System), Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - VA Puget Sound Health Care System, Seattle, Washington
  - West Virginia University Medicine, Morgantown, West Virginia
- Belgium (6):
  - AZ Sint-Lucas, Bruges
  - UZ Antwerp, Edegem
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - Jolimont Hospital, La Louvière
  - AZ Delta, Roeselare

REFERENCES:
- [Derived] Farsad K, Novelli PM, Laing C, Gandhi RT, Cynamon J, Lopez CS, Stempinski ES, Strasser R, Agah R. Double-Balloon Catheter-Mediated Transarterial Chemotherapy Delivery in a Swine Model: A Mechanism Recruiting the Vasa Vasorum for Localized Therapies. J Vasc Interv Radiol. 2024 Jul;35(7):1043-1048.e3. doi: 10.1016/j.jvir.2024.03.016. Epub 2024 Mar 18. PMID 38508449